CLINICAL TRIAL: NCT06495385
Title: Evaluation of a Multidisciplinary Care Pathway on the Evolution of Renal Function in Patients With Advanced Chronic Kidney Disease
Status: Active, not recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Other Study IDs: IRBN1502023/CHUSTE
Record Dates: First submitted 2024-01-26; First posted 2024-07-10 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-07

CONDITIONS: Chronic Kidney Disease stage4; Chronic Kidney Disease Stage 5
Keywords: Multidisciplinary Care; Pathway; Chronic Kidney disease; Patients' education
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Study group: Full participation (medical + dietitian+ specialist nurse)
  Interventions: Diagnostic Test: Evolution of renal function; Diagnostic Test: Measurement of haemoglobin levels; Diagnostic Test: Measurement of biological parameters; Diagnostic Test: Measure sodium and protein consumption; Behavioral: Quality of life questionnaire EUROQOL 5 dimensions (EQ-5D-5L)
- Control 1: Partial participation (medical+ dietitian OR specialist nurse)
  Interventions: Diagnostic Test: Evolution of renal function; Diagnostic Test: Measurement of haemoglobin levels; Diagnostic Test: Measurement of biological parameters; Diagnostic Test: Measure sodium and protein consumption; Behavioral: Quality of life questionnaire EUROQOL 5 dimensions (EQ-5D-5L)
- Control 2: No participation (medical visit only)
  Interventions: Diagnostic Test: Evolution of renal function; Diagnostic Test: Measurement of haemoglobin levels; Diagnostic Test: Measurement of biological parameters; Diagnostic Test: Measure sodium and protein consumption; Behavioral: Quality of life questionnaire EUROQOL 5 dimensions (EQ-5D-5L)

INTERVENTIONS:
Diagnostic Test: Evolution of renal function — Plasma creatinine levels and glomerular filtration rate estimated using the CKD-Epi formula adjusted for 1.73 m2 body surface area will be measured.
Diagnostic Test: Measurement of haemoglobin levels — Haemoglobin levels will be measured.
Diagnostic Test: Measurement of biological parameters — Plasma levels of urea, calcium, phosphorus and parathyroid hormone, as well as alkaline reserve, will be measured.
Diagnostic Test: Measure sodium and protein consumption — 24-hour urine volume, proteinuria, urea and sodium, will be measured.
Behavioral: Quality of life questionnaire EUROQOL 5 dimensions (EQ-5D-5L) — The descriptive system comprises five dimensions: mobility, personal care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, mild problems, moderate problems, severe problems and extreme problems. The figures for the five dimensions can be combined into a 5-digit number describing the patient's state of health. Scores close to 1 indicate "the best health you can imagine" and those close to 0 "the worst health you can imagine".

SUMMARY:
The number of incident and prevalent patients with end stage renal disease on dialysis treatment is increasing in France and worldwide. A quarter of dialysis patients are initiating dialysis urgently through central venous catheters and the number of patients registered in the waiting list for renal transplantation before dialysis initiation is very low. This is also reflected in the very low number of pre-emptive renal transplantations.

In order to reduce the number of dialysis patients, the French state has induced a national program proposing a multidisciplinary care pathway including the nephrology visits and at least one consultation with a dietitian and a specialist renal nurse in all patients with Chronic Kidney Disease stage 4 and 5.

DETAILED DESCRIPTION:
The aim of this single-center retrospective study is to evaluate the influence of the complete, partial or no participation in this program on the evolution of renal function and clinicobiological parameters in this group of patients.

ELIGIBILITY:
Inclusion Criteria:

* All stage 4 and 5 Chronic Kidney Disease patients that were included in the program from 01/01/2021 to 31/12/2021 in the clinics of AURA SANTE

Exclusion Criteria:

* Patients without a medical follow up during this year (2021)
* Patients with insufficient or no data during the 24 month of follow up period
* Active treatment with corticosteroids, cytotoxic or immunosuppressive drugs, ongoing infection, autoimmune disease or active tumor process.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with advanced chronic kidney disease will be included.
Sampling Method: Non-Probability Sample
Enrollment: 535 (Estimated)
Dates: Start 2024-04-09 (Actual); Primary Completion 2024-05-22 (Actual); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Evolution of estimated Glomerular filtration rate with the CKD-EPI formula adjusted for 1.73m2 of body surface area for the three groups | Month : 6, 12, 18 and 24
  The estimated Glomerular filtration rate is estimated with the CKD-EPI formula adjusted for 1.73m2 of body surface area and produced in ml/min/1.73m2 of body surface area. The CKD-EPI formula used is as follows: The conversion of serum creatinine level for the CKD-EPI formula was done as follows: creatinine level (mg/dl) = creatinine level (μmol/l) × 0.01131222 (considering that 1 mg/dl creatinine = 88.4 μmol/l creatinine). A GFR of 60 or more is within the normal range. A GFR below 60 may indicate kidney disease.

SECONDARY OUTCOMES:
Evolution of renal survival over the follow up period for every group | Month : 6, 12, 18 and 24
  Renal survival is measured as a percentage of remaining patients from baseline.
Evolution of patients' survival for every group during the study period | Month : 6, 12, 18 and 24
  Patients survival is measured as a percentage of remaining patients from baseline.
Evolution of preemptive transplantation during the study period for the three study groups | Month : 6, 12, 18 and 24
  The number of preventive transplants will be compared in each group.
Evolution of biological parameters : Haemoglobin | Month : 6, 12, 18 and 24
  Haemoglobin levels are measured as gram/dL.
Evolution of biological parameters : plasma calcium | Month : 6, 12, 18 and 24
  Plasma Calcium levels are measured as mg/dL.
Evolution of biological parameters : phosphate | Month : 6, 12, 18 and 24
  Plasma Phosphate levels are measured as mg/dL.
Evolution of biological parameters : parathyroid hormone | Month : 6, 12, 18 and 24
  Plasma parathyroid hormone levels are measured in pg/ml.
Evolution of biological parameters : alkaline reserve levels | Month : 6, 12, 18 and 24
  Plasma alkaline reserve levels are measured in mmol/l.
Evolution of dietary parameters : salt consumption | Month : 6, 12, 18 and 24
  24h salt consumption are measured in g/24h.
Evolution of dietary parameters : protein consumption | Month : 6, 12, 18 and 24
  24h protein consumption are measured in g/24h.
Quality of life questionnaire EUROQOL 5 dimensions (EQ-5D-5L) | Month : 6, 12, 18 and 24
  The descriptive system comprises five dimensions: mobility, personal care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, mild problems, moderate problems, severe problems and extreme problems. The figures for the five dimensions can be combined into a 5-digit number describing the patient's state of health. Scores close to 1 indicate "the best health you can imagine" and those close to 0 "the worst health you can imagine".

CONTACTS AND LOCATIONS:
Overall Officials: Hélène PAGES, nurse, Principal Investigator — CHU de Saint-Etienne
Locations (1):
- AURA Santé, Chamalières, France

IPD SHARING:
Plan to Share IPD: No